CLINICAL TRIAL: NCT01000298
Title: Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Effectiveness of Oral Antibiotics in the Community-based Treatment of Severe Acute Malnutrition in Malawian Children
Brief Title: Effectiveness of Oral Antibiotics in the Treatment of Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Professor Mark J. Manary, Washington Univeristy in St. Louis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJM-antibiotics
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Kwashiorkor; Marasmus
MeSH Terms: conditions — Kwashiorkor; Protein-Energy Malnutrition | interventions — Amoxicillin; Cefdinir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Amoxicillin (Experimental)
  Interventions: Drug: Amoxicillin
- cefdinir (Experimental): cefdinir
  Interventions: Drug: Cefdinir

INTERVENTIONS:
Drug: Placebo — liquid placebo medication given twice per day for 7 days
  Arms: Placebo
Drug: Amoxicillin — liquid amoxicillin given twice per day for 7 days
  Arms: Amoxicillin
Drug: Cefdinir — liquid cefdinir given twice per day for 7 days
  Other Names: Omnicef
  Arms: cefdinir

SUMMARY:
The need for oral antibiotics as part of the case management of severe acute malnutrition (SAM) in the outpatient setting has not been studied in a prospective trial. This study will compare the recovery rates of children with SAM treated at home with locally-produced ready-to-use therapeutic food (RUTF) with and without prescribed antibiotics as part of their outpatient case management. The investigators hypothesize that there will be no significant difference in rates of recovery between children who receive and children who do not receive antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* 6 months - 5 years old
* Kwashiorkor or Marasmus
* Qualifies for home-based therapeutic feeding with RUTF

Exclusion Criteria:

* Obvious congenital or other malformation that makes child a poor candidate for home-based feeding with RUTF
* Unable to consume test-dose of RUTF in clinic
* Parent refusal to participate and return for follow-up

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2700 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
nutritional recovery | 12 weeks

SECONDARY OUTCOMES:
weight gain | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Nutrition Project, Blantyre, Malawi

REFERENCES:
- [Derived] Trehan I, Goldbach HS, LaGrone LN, Meuli GJ, Wang RJ, Maleta KM, Manary MJ. Antibiotics as part of the management of severe acute malnutrition. Malawi Med J. 2016 Sep;28(3):123-130. PMID 27895846
- [Derived] Trehan I, Goldbach HS, LaGrone LN, Meuli GJ, Wang RJ, Maleta KM, Manary MJ. Antibiotics as part of the management of severe acute malnutrition. N Engl J Med. 2013 Jan 31;368(5):425-35. doi: 10.1056/NEJMoa1202851. PMID 23363496